CLINICAL TRIAL: NCT01379274
Title: A Phase II Trial of Revlimid® (Lenalidomide) and Low Dose Vidaza® (Azacitidine) in Patients With Low - Intermediate-1 Risk Myelodysplastic Syndromes
Brief Title: A Trial of Lenalidomide & Azacitidine in Low Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: Rush University Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Jamile Shammo, Associate Professor of Medicine and Pathology, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS 2008-01
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: MDS
Keywords: MDS; Low risk disease; IPSS
MeSH Terms: interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide and azacitidine combination (Experimental): Lenalidomide and azacitidine combination to be utilized in patients who did not respond to 3 months of lenalidomide monotherapy.
  Interventions: Drug: Lenalidomide and azacitidine combination

INTERVENTIONS:
Drug: Lenalidomide and azacitidine combination — lenalidomide 10 mg will be administered orally on Days 1-28 of each 28-day cycle. Patients who fail to achieve an erythroid response per 2006 IWG criteria after 3 cycles of monotherapy will receive lenalidomide at the same dose administered in cycle 3 and low-dose azacitidine25 mg/m2 subcutaneously (SC) or intravenously (IV) for 5 days (on Days 1-5) of every 28-day cycle.
  Patients who fail to respond (2006 IWG criteria) after receiving two cycles of combination therapy will receive lenalidomide at the same dose administered in Cycle 3 and azacitidine 50 mg/m2 SC or IV given daily on Days 1-5 of each 28-day cycle, if no grade 4 toxicity developed or no delay greater than 2 weeks in starting a new cycle was experienced during the first 2 cycles of combination therapy.
  Other Names: lenalidomide; Azacitidine

SUMMARY:
This phase II study will evaluate the safety and efficacy of combining two active agents;Revlimid® (lenalidomide) and low dose Vidaza® (azacitidine) for the treatment of patients with low to intermediate-1 MDS excluding patients with 5 q deletion. The rationale for adding Vidaza® (azacitidine) after 3 months of revlimid monotherapy is that combination therapy will result in higher response rates, and potentially longer response duration than that achieved with either agent.

STUDY OBJECTIVES:

Primary:

To determine the safety and tolerability of the combination of Revlimid® (lenalidomide) and low dose Vidaza® (azacitidine) in patients with low - intermediate-1 risk MDS non 5 q deletion who have not responded after 3 months of Revlimid® (lenalidomide) monotherapy

Secondary:

To determine the response rate in patients with low - intermediate-1 risk MDS non 5 q deletion receiving Revlimid® (lenalidomide) in combination with low dose Vidaza® (azacitidine), as defined by the IWG 2006 Revised Response Criteria

DETAILED DESCRIPTION:
Eligibility criteria

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosis of low- or intermediate-1-risk IPSS (see Appendix III) MDS without an abnormality of chromosome 5 involving a deletion between bands q31 and q33.

   Pathologic diagnosis via pathology performed at Rush University Medical Center or made available to Rush from outside institution.
5. Prior treatment with < 3 cycles (84 days) of Revlimid® (lenalidomide) are eligible for enrollment regardless of response.
6. ECOG performance status of 2 at study entry (see Appendix II).
7. Disease free of prior malignancies for > 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
8. Serum bilirubin levels < 1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
9. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels < 2 x ULN.
10. Serum creatinine levels < 1.5 x ULN
11. Absolute neutrophil count > 1000/mm³
12. Platelet count > 30,000/mm³
13. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

ELIGIBILITY:
Inclusion Criteria: Patients with low to Int-1 risk MDS

1. ECOG performance status of < 2 at study entry (see Appendix II).
2. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
3. Serum bilirubin levels < 1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
4. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels < 2 x ULN.
5. Serum creatinine levels 1.5 x ULN
6. Absolute neutrophil count > 1000/mm³
7. Platelet count > 30,000/mm³
8. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
9. Females of childbearing potential (FCBP)† must have a negative serum or urine

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. Lactating females must agree not to breast feed while taking Revlimid® (lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to lenalidomide, azacitidine, or mannitol.
6. Any prior use of Vidaza® (azacitidine).
7. Prior use of Revlimid® (lenalidomide) for more than 84 days (three 28 day cycles).
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or infectious hepatitis, type B or C.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamile M Shammo, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from approximately 2010-2012.
Groups:
- Lenalidomide and Azacitidine Combination: Lenalidomide and azacitidine combination to be utilized in patients who did not respond to 3 months of lenalidomide monotherapy.
  Lenalidomide and azacitidine combination: lenalidomide 10 mg will be administered orally on Days 1-28 of each 28-day cycle. Patients who fail to achieve an erythroid response per 2006 IWG criteria after 3 cycles of monotherapy will receive lenalidomide at the same dose administered in cycle 3 and low-dose azacitidine25 mg/m2 subcutaneously (SC) or intravenously (IV) for 5 days (on Days 1-5) of every 28-day cycle.
  Patients who fail to respond (2006 IWG criteria) after receiving two cycles of combination therapy will receive lenalidomide at the same dose administered in Cycle 3 and azacitidine 50 mg/m2 SC or IV given daily on Days 1-5 of each 28-day cycle, if no grade 4 toxicity developed or no delay greater than 2 weeks in starting a new cycle was experienced during the first 2 cycles of combination therapy.
Period: Overall Study
Arm/Group | Lenalidomide and Azacitidine Combination
Started | 2
Completed | 1
Not Completed | 1
Not completed — funding withdrawn | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and Azacitidine Combination
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Revlimid and Azacitidine Combination
Description: To determine the number of subjects who develop grade 4 toxicity while on combination therapy.
Time Frame: Study was closed and outcome unable to be measured.
Population: Study was unable to be completed since funding was withdrawn.
Arm/Group | Lenalidomide and Azacitidine Combination
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study ended early. Data not analyzed.
Description: Study ended early. Data not analyzed.
Arm/Group | Lenalidomide and Azacitidine Combination
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study was not able to be completed since funding was withdrawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No